CLINICAL TRIAL: NCT02470481
Title: Psoriatic Arthritis In Skin Clinics (PARIS) Study. A Multicentre, Observational, Descriptive Cross-Cultural Validation Study and Estimate of the Proportion of Patients With Psoriatic Arthritis Among Psoriasis Patients Attending Dermatology Clinics Selected for This Study
Brief Title: A Study in Participants With Psoriatic Arthritis Attending Dermatology Clinics
Acronym: PARIS
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR103908; CNTO148PSA4001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-06-10; First posted 2015-06-12 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: Participants with psoriatic arthritis among psoriasis particiants attending dermatology clinics.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is an obervational study

SUMMARY:
The purpose of this study is to conduct full psychometric testing of the Early Arthritis for Psoriatic Patients (EARP) questionnaire in Australian, Korean and Chinese populations

DETAILED DESCRIPTION:
This is a multicentre, observational, descriptive estimate of the proportion of participants with psoriatic arthritis among psoriasis participants attending dermatology clinics selected for this study. In addition, this study will involve full psychometric assessment of the Early psoriatic screening questionnaire (EARP) questionnaire with the aim of identifying and appropriately referring participants to a rheumatologist for review if their EARP score is 3 or greater at Screening (i.e. >= 3 at Visit 1).

ELIGIBILITY:
Inclusion Criteria:

* Patient must be a man or woman aged 18 to 65 years of age, inclusive
* The patient must have an established diagnosis of psoriasis (based upon clinical evidence, and documented medical history [19])
* The patient must be able to read and write in the target language (English, Mandarin or Korean; or other relevant target languages)
* Each patient must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* An established diagnosis of psoriatic arthritis
* Ever have received systemic treatment with a disease modifying antirheumatic drug (DMARD) for arthritis or spondylitis (inflammatory back pain)
* Ever have received systemic treatment with a biologic therapy for psoriasis (including infliximab, golimumab, ustekinumab, adalimumab or etanercept)
* A history of employment in or are currently employed in the healthcare industry; or
* Participated in the translation and linguistic validation of the EARP questionnaire

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with psoriatic arthritis among psoriasis participants attending dermatology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2015-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Psoriatic Arthritis | Baseline up to Day 28
  Percentage of participants with psoriatic arthritis will be assessed using formula: Number of participants diagnosed with psoriatic arthritis divided by total number of participants with psoriasis attending the dermatology clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (5):
- Australia (2):
  - Fitzroy
  - New Lambton
- China (2):
  - Beijing
  - Hangzhou
- Seoul, South Korea

REFERENCES:
- [Derived] Jo SJ, Foley P, Oakley SP, Zhang J, Zheng M, Shin K, McGonagle D, Gisondi P, Tinazzi I, Butcher BE, Handel M. Initial assessment of the early arthritis for psoriatic patients diagnostic questionnaire in dermatology clinics in Australia, Korea and China. Int J Rheum Dis. 2019 Aug;22(8):1512-1520. doi: 10.1111/1756-185X.13604. Epub 2019 May 22. PMID 31115158